CLINICAL TRIAL: NCT04380389
Title: Accuracy of ScanWatch Pulse Oximeter With Profound Hypoxia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Withings (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: pulse ox
Record Dates: First submitted 2020-05-05; First posted 2020-05-08 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Oximetry

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- profound hypoxia (Other)
  Interventions: Diagnostic Test: hypoxia

INTERVENTIONS:
Diagnostic Test: hypoxia — Brief stable arterial oxygen desaturation in healthy volunteers and sampling arterial blood when a stable level of hypoxia has been attained.

SUMMARY:
Performance testing of pulse oximeters. The protocol involves brief stable arterial oxygen desaturation in healthy volunteers and sampling arterial blood when a stable level of hypoxia has been attained. The blood sample is analyzed for oxygen saturation with a gold standard bench CO-oximeter. This protocol is aligned with the latest ISO and FDA guidance documents for pulse oximeter testing.

ELIGIBILITY:
Inclusion Criteria:

* The subject is male or female, aged ≥18 and <50.
* The subject is in good general health with no evidence of any medical problems.
* The subject has both wrist circumferences between 14 and 22cm.
* The subject has provided informed consent and is willing to comply with the study procedures.

Exclusion Criteria:

* The subject is obese (BMI>30).
* The subject has a known history of heart disease, lung disease, kidney or liver disease.
* Diagnosis of asthma, sleep apnea, or use of CPAP.
* Subject has diabetes.
* Subject has a clotting disorder.
* The subject a hemoglobinopathy or history of anemia, per subject report or the first blood sample that in the opinion of the investigator, would make them unsuitable for study participation.
* The subject has any other serious systemic illness.
* The subject is a current smoker.
* The subject has piercings that may cause air leaks during the test
* The subject has any injury, deformity, or abnormality at the sensor sites that in the opinion of the investigators' would interfere with the sensors working correctly.
* The subject has a history of fainting or vasovagal response.
* The subject has a history of sensitivity to local anesthesia.
* The subject has a diagnosis of Raynaud's disease.
* The subject has unacceptable collateral circulation based on exam by the investigator (Allen's test).
* The subject is pregnant, lactating or trying to get pregnant.
* The subject is unable or unwilling to provide informed consent, or is unable or unwilling to comply with study procedures.
* The subject has a resting heartrate over 120, Systolic BP is over 150, diastolic BP is over 90 or room air SpO2 is less than 94%.
* The subject has carboxyhemoglobin over 3% as measured by Lab blood gas analysis.
* The subject has any other condition, which in the opinion of the investigators' would make them unsuitable to participate.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2020-03-11 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
RMSE compared to CO-oximetry | 1 hour
  Root Mean Squared Error between the functional blood oxygen saturation (SpO2) provided by the device under test and the arterial blood oxygen measured with the CO-oximeter.

CONTACTS AND LOCATIONS:
Locations (1):
- Hypoxia Lab, UCSF, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kirszenblat R, Edouard P. Validation of the Withings ScanWatch as a Wrist-Worn Reflective Pulse Oximeter: Prospective Interventional Clinical Study. J Med Internet Res. 2021 Apr 26;23(4):e27503. doi: 10.2196/27503. PMID 33857011
- See also: Pulse Oximeters - Premarket Notification Submissions [510(k)s] Guidance for Industry and Food and Drug Administration Staff, March 4, 2013 — https://www.fda.gov/regulatory-information/search-fda-guidance-documents/pulse-oximeters-premarket-notification-submissions-510ks-guidance-industry-and-food-and-drug
- See also: ISO 80601-2-61:2017 Medical electrical equipment - Part 2-61: Particular requirements for basic safety and essential performance of pulse oximeter equipment — https://www.iso.org/fr/standard/67963.html